CLINICAL TRIAL: NCT01711892
Title: A Randomized Controlled Clinical Trial on the Effects of Recreational Soccer Training in Men With Prostate Cancer Receiving Androgen Deprivation Therapy: The FC Prostate Study
Brief Title: Health Effects of Soccer Training in Men With Prostate Cancer Receiving Androgen Deprivation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Danish Cancer Society (Other); Novo Nordisk A/S (Industry); TrygFonden, Denmark (Industry); Beckett Foundation (Other)
Responsible Party: Principal Investigator, Jacob Uth, Project manager, Ph.d student, Master of Health Science, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CIRE-04
Record Dates: First submitted 2012-10-17; First posted 2012-10-22 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Prostatic Neoplasms; Exercise; Soccer Training; Androgen Deprivation Therapy
Keywords: Prostatic Neoplasms; Prostate Cancer; Exercise; Soccer; Androgen Deprivation Therapy; Body Composition; Cardiovascular fitness; Bone Health; Health Related Quality of Life
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Soccer Training (Active Comparator): 12 weeks of soccer training. (2 times per week for the first 8 weeks and 3 times per week in the last 4 weeks. Training will consist of 15 minutes warm-up and 2 x 15 minutes matches for the first 4 weeks and of 15 minutes warm-up and 3 x 15 minutes matches for the last 8 weeks). After 12 weeks assessments participants in the intervention group will continue bi-weekly supervised training for additional 20 weeks at the end of which tests will be repeated.
  Interventions: Behavioral: Soccer training
- Control group (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Soccer training
  Arms: Soccer Training

SUMMARY:
Androgen Deprivation Therapy (ADT) is standard treatment for locally advanced or advanced Prostate Cancer (PC).

The musculoskeletal toxicity associated with ADT is well established, leading to a decrease in muscle mass, increased fat percentage, weight gain, sexual dysfunction and increased risk of depression, fatigue, diabetes, cardiovascular disease and reduced quality of life.

Numerous studies have shown an association between physical activity, physical capacity and quality of life in cancer patients and recent epidemiological research suggest that regular, moderate-intensity physical activity may have a positive effect on survival in men with prostate cancer.

Within exercise physiology there is new evidence pointing to recreational soccer as a unique form of intermittent exercise that effectively stimulates aerobic and anaerobic energy delivery systems, leading to beneficial musculoskeletal, metabolic and cardiovascular adaptations of importance for health.

It is our overall hypothesis that 12 weeks of recreational soccer training 2-3 times per week will improve the health profile of PC patients receiving ADT treatment.

ELIGIBILITY:
Inclusion Criteria:

- Patients with locally advanced or advanced prostate cancer being treated with androgen deprivation therapy (S-testosterone < 1.7) for at least 6 months at the time of inclusion

Exclusion Criteria:

* WHO performance level above 1,symptomatic cardiovascular disorders, osteoporosis (T-score below -2.5)

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2012-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Baseline to post intervention (12 weeks) and follow-up (32 weeks) change in Body Composition. | Change from baseline to post intervention (12 weeks) and follow-up (32 weeks)
  Changes in body composition assessed by Dual-energy X-ray absorptiometry(DXA)scan

SECONDARY OUTCOMES:
Bone Mineral Density | Change from baseline to post intervention (12 weeks) and follow-up (32 weeks)
Cardiorespiratory fitness (Vo2 peak) | Change from baseline to post intervention (12 weeks) and follow-up (32 weeks)
  Change in maximal oxygen consumption (Vo2 peak) assessed directly during an incremental test on a cycle ergometer from baseline to post-intervention (12 weeks) and follow-up (32 weeks).
Patient reported outcomes | Change from baseline to post intervention (12 weeks) and follow-up (32 weeks)
  Changes in Psychological distress (Hospital Anxiety and Depression Scale, HADS), Quality of Life (EORTC QLQ C-30), general well-being (SF-36), disease specific symptoms and side-effects (EORTC PR-25)from baseline to post-intervention (12 weeks) and follow-up (32 weeks)
Heart function | Change from baseline to post intervention (12 weeks) and follow-up (32 weeks)
  Changes in Heart function measured by Echocardiography from baseline to post-intervention (12 weeks) and follow-up (32 weeks)
Glucose tolerance | Change from baseline to post intervention (12 weeks) and follow-up (32 weeks)
  Oral Glucose Tolerance Test
Postural Balance | Change from baseline to post intervention (12 weeks) and follow-up (32 weeks)
  Assessed standing on a force platform with feet in bilateral, unilateral and tandem position. Additionally assessed with a modified Flamingo balance test.
Physical function | Change from baseline to post intervention (12 weeks) and follow-up (32 weeks)
  Physical function will be assessed with sit to stand test (30s), stair climbing test and Counter Movement Jump (jump height)
Hip to waist ratio | Change from baseline to post intervention (12 weeks) and follow-up (32 weeks)
  Hip and waist circumference will be measured and the hip to waist ratio will be calculated
Muscle Strength | Change from baseline to post intervention (12 weeks) and follow-up (32 weeks)
  Muscle strength will be assessed with the 1Repetition Maximum test for knee extensors
Blood markers | Change from baseline to post intervention (12 weeks) and follow-up (32 weeks)
  Markers of inflammation and bone metabolism will be obtained after overnight fasting

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Rørth, Professor, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Centre of Integrated Rehabilitation of Cancer Patients, Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Uth J, Hornstrup T, Christensen JF, Christensen KB, Jorgensen NR, Helge EW, Schmidt JF, Brasso K, Helge JW, Jakobsen MD, Andersen LL, Rorth M, Midtgaard J, Krustrup P. Football training in men with prostate cancer undergoing androgen deprivation therapy: activity profile and short-term skeletal and postural balance adaptations. Eur J Appl Physiol. 2016 Mar;116(3):471-80. doi: 10.1007/s00421-015-3301-y. Epub 2015 Nov 30. PMID 26620651
- [Derived] Uth J, Hornstrup T, Christensen JF, Christensen KB, Jorgensen NR, Schmidt JF, Brasso K, Jakobsen MD, Sundstrup E, Andersen LL, Rorth M, Midtgaard J, Krustrup P, Helge EW. Efficacy of recreational football on bone health, body composition, and physical functioning in men with prostate cancer undergoing androgen deprivation therapy: 32-week follow-up of the FC prostate randomised controlled trial. Osteoporos Int. 2016 Apr;27(4):1507-1518. doi: 10.1007/s00198-015-3399-0. Epub 2015 Nov 16. PMID 26572756
- [Derived] Bruun DM, Krustrup P, Hornstrup T, Uth J, Brasso K, Rorth M, Christensen JF, Midtgaard J. "All boys and men can play football": a qualitative investigation of recreational football in prostate cancer patients. Scand J Med Sci Sports. 2014 Aug;24 Suppl 1:113-21. doi: 10.1111/sms.12193. PMID 24944135
- [Derived] Uth J, Hornstrup T, Schmidt JF, Christensen JF, Frandsen C, Christensen KB, Helge EW, Brasso K, Rorth M, Midtgaard J, Krustrup P. Football training improves lean body mass in men with prostate cancer undergoing androgen deprivation therapy. Scand J Med Sci Sports. 2014 Aug;24 Suppl 1:105-12. doi: 10.1111/sms.12260. PMID 24944134
- [Derived] Krustrup P, Hansen PR, Nielsen CM, Larsen MN, Randers MB, Manniche V, Hansen L, Dvorak J, Bangsbo J. Structural and functional cardiac adaptations to a 10-week school-based football intervention for 9-10-year-old children. Scand J Med Sci Sports. 2014 Aug;24 Suppl 1:4-9. doi: 10.1111/sms.12277. PMID 24944128
- [Derived] Uth J, Schmidt JF, Christensen JF, Hornstrup T, Andersen LJ, Hansen PR, Christensen KB, Andersen LL, Helge EW, Brasso K, Rorth M, Krustrup P, Midtgaard J. Effects of recreational soccer in men with prostate cancer undergoing androgen deprivation therapy: study protocol for the 'FC Prostate' randomized controlled trial. BMC Cancer. 2013 Dec 13;13:595. doi: 10.1186/1471-2407-13-595. PMID 24330570